CLINICAL TRIAL: NCT03054025
Title: Facilitating Motivational Readiness and Adoption of Physical Activity by Breast Cancer Survivors With a Smart Phone Application
Brief Title: Smart Phone Application in Increasing Physical Activity in Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding discontinued
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15G.393; JT 7946 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (smart phone application) (Experimental): Participants download the physical activity readiness smart phone application onto their personal smartphone and receive training on how to use the app which includes animated video clips, tailored email reminders, and feedback on progress for 3 weeks.
  Interventions: Device: Smart Phone Monitoring Device

INTERVENTIONS:
Device: Smart Phone Monitoring Device — Use activity tracker application
  Other Names: Monitor

SUMMARY:
This pilot clinical trial studies how well a smart phone application works in increasing physical activity in breast cancer survivors. A smart phone application that increases physical activity may help reduce the likelihood of cancer coming back in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a pilot study to inform the design of a mobile health application for smartphone that is targeted to increase physical activity and reduce risks associated with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* A participant is only able to participate in one phase, not both phases, of the research study
* Must have completed breast cancer treatment
* Those on adjuvant hormonal therapy are allowed to participate in the research study (either phase)

Exclusion Criteria:

* Those who currently meet the Centers for Disease Control and Prevention (CDC)'s physical activity guidelines
* Those who do not currently use a smartphone (of any kind)
* Those who do not read and speak English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Features of the mobile application that were most used by participants | 3 weeks
  Descriptive statistics using proportions and 90% confidence intervals will be calculated for various features.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Barsevick, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/